CLINICAL TRIAL: NCT01155726
Title: The Effect of Masking on Subjective Results During Daily Disposable Contact Lens Studies
Acronym: ARGON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIBA VISION (Industry)
Responsible Party: Sponsor
Organization: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P-371-C-101
Record Dates: First submitted 2010-06-30; First posted 2010-07-02 (Estimated); Results first posted 2012-05-15 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-04

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia | interventions — Masks

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nelfilcon A, Masked, Unmasked (Active Comparator): Nelfilcon A worn in adaptation phase (bilaterally, 30 days). Period 1: 1DAVM and DACP (masked) worn contralaterally in random assignment for 3 days. Period 2: 1DAVM and DACP (unmasked) worn contralaterally, same assignment, 3 days. All products worn in a daily wear, daily disposable mode.
  Interventions: Device: Nelfilcon A contact lens; Device: Nelfilcon A contact lens with comfort additive (DACP), unmasked; Device: Nelfilcon A contact lens with comfort additive (DACP), masked; Device: Etafilcon A contact lens with comfort additive (1DAVM), unmasked; Device: Etafilcon A contact lens with comfort additive (1DAVM), masked
- Nelfilcon A, Masked, Partially Masked (Active Comparator): Nelfilcon A worn in adaptation phase (bilaterally, 30 days). Period 1: 1DAVM and DACP (masked) worn contralaterally in random assignment for 3 days. Period 2: 1DAVM and DACP (partially masked) worn contralaterally, same assignment, 3 days. All products worn in a daily wear, daily disposable mode.
  Interventions: Device: Nelfilcon A contact lens; Device: Nelfilcon A contact lens with comfort additive (DACP), masked; Device: Nelfilcon A contact lens with comfort additive (DACP), partially masked; Device: Etafilcon A contact lens with comfort additive (1DAVM), masked; Device: Etafilcon A contact lens with comfort additive (1DAVM), partially masked
- Etafilcon A, Masked, Unmasked (Active Comparator): Etafilcon A worn in adaptation phase (bilaterally, 30 days). Period 1: 1DAVM and DACP (masked) worn contralaterally in random assignment for 3 days. Period 2: 1DAVM and DACP (unmasked) worn contralaterally, same assignment, 3 days. All products worn in a daily wear, daily disposable mode.
  Interventions: Device: Nelfilcon A contact lens with comfort additive (DACP), unmasked; Device: Nelfilcon A contact lens with comfort additive (DACP), masked; Device: Etafilcon A contact lens; Device: Etafilcon A contact lens with comfort additive (1DAVM), unmasked; Device: Etafilcon A contact lens with comfort additive (1DAVM), masked
- Etafilcon A, Masked, Partially Masked (Active Comparator): Etafilcon A worn in adaptation phase (bilaterally, 30 days). Period 1: 1DAVM and DACP (masked) worn contralaterally in random assignment for 3 days. Period 2: 1DAVM and DACP (partially masked) worn contralaterally, same assignment, 3 days. All products worn in a daily wear, daily disposable mode.
  Interventions: Device: Nelfilcon A contact lens with comfort additive (DACP), masked; Device: Nelfilcon A contact lens with comfort additive (DACP), partially masked; Device: Etafilcon A contact lens; Device: Etafilcon A contact lens with comfort additive (1DAVM), masked; Device: Etafilcon A contact lens with comfort additive (1DAVM), partially masked

INTERVENTIONS:
Device: Nelfilcon A contact lens — Commercially marketed, soft, hydrogel contact lens for daily wear, daily disposable use. Blister pack label and lens packaging visible to participant. Lenses inserted and removed by participant.
  Other Names: Focus DAILIES®
  Arms: Nelfilcon A, Masked, Partially Masked; Nelfilcon A, Masked, Unmasked
Device: Nelfilcon A contact lens with comfort additive (DACP), unmasked — Commercially marketed, soft, hydrogel contact lens with comfort additive for daily wear, daily disposable use. Blister pack label and lens packaging visible to participant. Lenses and removed inserted by participant.
  Other Names: DAILIES® AquaComfort Plus®
  Arms: Etafilcon A, Masked, Unmasked; Nelfilcon A, Masked, Unmasked
Device: Nelfilcon A contact lens with comfort additive (DACP), masked — Commercially marketed, soft, hydrogel contact lens for daily wear, daily disposable use. Blister pack label and packaging not visible to participant. Lenses inserted and removed by the investigator.
  Other Names: DAILIES® AquaComfort Plus®
Device: Nelfilcon A contact lens with comfort additive (DACP), partially masked — Commercially marketed, soft, hydrogel contact lens for daily wear, daily disposable use. Lens name and manufacturer on blister pack label concealed from participant. Lenses inserted and removed by the participant.
  Other Names: DAILIES® AquaComfort Plus®
  Arms: Etafilcon A, Masked, Partially Masked; Nelfilcon A, Masked, Partially Masked
Device: Etafilcon A contact lens — Commercially marketed, soft, hydrogel contact lens for daily wear, daily disposable use. Blister pack label and lens packaging visible to participant. Lenses inserted and removed by participant.
  Other Names: 1-DAY ACUVUE®
  Arms: Etafilcon A, Masked, Partially Masked; Etafilcon A, Masked, Unmasked
Device: Etafilcon A contact lens with comfort additive (1DAVM), unmasked — Commercially marketed, soft, hydrogel contact lens with comfort additive for daily wear, daily disposable use. Blister pack label and lens packaging visible to participant. Lenses inserted and removed by participant.
  Other Names: 1-DAY ACUVUE® MOIST®
  Arms: Etafilcon A, Masked, Unmasked; Nelfilcon A, Masked, Unmasked
Device: Etafilcon A contact lens with comfort additive (1DAVM), masked — Commercially marketed, soft, hydrogel contact lens for daily wear, daily disposable use. Blister pack label and packaging not visible to participant. Lenses inserted and removed by the investigator.
  Other Names: 1-DAY ACUVUE® MOIST®
Device: Etafilcon A contact lens with comfort additive (1DAVM), partially masked — Commercially marketed, soft, hydrogel contact lens for daily wear, daily disposable use. Lens name and manufacturer on blister pack label concealed from participant. Lenses inserted and removed by the participant.
  Other Names: 1-DAY ACUVUE® MOIST®
  Arms: Etafilcon A, Masked, Partially Masked; Nelfilcon A, Masked, Partially Masked

SUMMARY:
The purpose of this study is to explore the effect of masking on subjective ratings for two daily disposable contact lenses.

ELIGIBILITY:
Inclusion Criteria:

* 17 years of age or older.
* Ocular exam within 2 years.
* Currently wearing soft contact lenses on a daily wear basis.
* Contact lens prescription between +6.00D and -10.00D.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any ocular disease.
* Use of systemic or ocular medications that may affect ocular health.
* Unable to achieve an acceptable fit with the study lenses.
* Anisometropia >1.00D or astigmatism >0.75D.
* Other protocol-defined exclusion criteria may apply.

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Contact Lens Research: University of Waterloo, Waterloo, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 134 participants were recruited and enrolled at 1 study center located in Canada. A 24-hour washout period of no lens wear preceded the 30-day adaptation phase.
Pre-assignment Details: 18 participants were enrolled but not dispensed--i.e., discontinued prior to the 30-day adaptation phase. 116 participants started the adaptation phase, and baseline characteristics are presented for this group. 2 discontinued during the adaptation phase and 15 discontinued between adaptation and Period 1 dispense. 99 were dispensed into Period 1.
Groups:
- Nelfilcon A, Masked, Unmasked: Nelfilcon A in adaptation phase. 1DAVM and DACP (contralateral wear, masked) in Period 1. 1DAVM and DACP (contralateral wear, unmasked) in Period 2.
- Nelfilcon A, Masked, Partially Masked: Nelfilcon A in adaptation phase. 1DAVM and DACP (contralateral wear, masked) in Period 1. 1DAVM and DACP (contralateral wear, partially masked) in Period 2.
- Etafilcon A, Masked, Unmasked: Etafilcon A in adaptation phase. 1DAVM and DACP (contralateral wear, masked) in Period 1. 1DAVM and DACP (contralateral wear, unmasked) in Period 2.
- Etafilcon A, Masked, Partially Masked: Etafilcon A in adaptation phase. 1DAVM and DACP (contralateral wear, masked) in Period 1. 1DAVM and DACP (contralateral wear, partially masked) in Period 2.
Period: Period 1, 3 Days (Masked)
Arm/Group | Nelfilcon A, Masked, Unmasked | Nelfilcon A, Masked, Partially Masked | Etafilcon A, Masked, Unmasked | Etafilcon A, Masked, Partially Masked
Started | 24 | 20 | 30 | 25
Completed | 23 | 20 | 28 | 25
Not Completed | 1 | 0 | 2 | 0
Not completed — Inconvenience | 1 | 0 | 2 | 0
Period: Period 2, 3 Days (Unmask) or (Partial)
Arm/Group | Nelfilcon A, Masked, Unmasked | Nelfilcon A, Masked, Partially Masked | Etafilcon A, Masked, Unmasked | Etafilcon A, Masked, Partially Masked
Started | 23 | 20 | 28 | 25
Completed | 23 | 20 | 28 | 25
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall: This reporting group includes all enrolled and dispensed participants.
Arm/Group | Overall
Number analyzed (Participants) | 116
Age Continuous [Mean (Standard Deviation); unit: years] | 25 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 37

OUTCOME MEASURES:

1. Primary Outcome: Average Subjective Comfort
Description: Participants were asked, "How would you rate your comfort with your study lenses?" and indicated their response by marking a continuum line ranging from 0=very poor comfort to 100=excellent comfort. Subjective comfort was collected at three time points (insertion, 4 hours, 8 hours) for 3 days, and the comfort ratings were averaged together.
Time Frame: Insertion, 4 hours, 8 hours each: Day 1, Day 2, and Day 3
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Nelfilcon A, Pd 1 Masked (1DAVM), Pd 2 Unmasked; Nelfilcon A, Pd 1 Masked (DACP), Pd 2 Unmasked; Nelfilcon A, Pd 1 Masked, Pd 2 Unmasked (1DAVM); Nelfilcon A, Pd 1 Masked, Pd 2 Unmasked (DACP): Nelfilcon A (adaptation phase), followed by Period 1 masked, Period 2 unmasked. Contralateral wear reported by product/eye.
- Etafilcon A, Pd 1 Masked (1DAVM), Pd 2 Unmasked; Etafilcon A, Pd 1 Masked (DACP), Pd 2 Unmasked; Etafilcon A, Pd 1 Masked, Pd 2 Unmasked (1DAVM); Etafilcon A, Pd 1 Masked, Pd 2 Unmasked (DACP): Etafilcon A (adaptation phase), followed by Period 1 masked, Period 2 unmasked. Contralateral wear reported by product/eye.
- Nelfilcon A, Pd 1 Masked (1DAVM), Pd 2 Partial; Nelfilcon A, Pd 1 Masked (DACP), Pd 2 Partial; Nelfilcon A, Pd 1 Masked, Pd 2 Partial (1DAVM); Nelfilcon A, Pd 1 Masked, Pd 2 Partial (DACP): Nelfilcon A (adaptation phase), followed by Period 1 masked, Period 2 partial masked. Contralateral wear reported by product/eye.
- Etafilcon A, Pd 1 Masked (1DAVM), Pd 2 Partial; Etafilcon A, Pd 1 Masked (DACP), Pd 2 Partial; Etafilcon A, Pd 1 Masked, Pd 2 Partial (1DAVM); Etafilcon A, Pd 1 Masked, Pd 2 Partial (DACP): Etafilcon A (adaptation phase), followed by Period 1 masked, Period 2 partial masked. Contralateral wear reported by product/eye.
Arm/Group | Nelfilcon A, Pd 1 Masked (1DAVM), Pd 2 Unmasked | Nelfilcon A, Pd 1 Masked (DACP), Pd 2 Unmasked | Etafilcon A, Pd 1 Masked (1DAVM), Pd 2 Unmasked | Etafilcon A, Pd 1 Masked (DACP), Pd 2 Unmasked | Nelfilcon A, Pd 1 Masked, Pd 2 Unmasked (1DAVM) | Nelfilcon A, Pd 1 Masked, Pd 2 Unmasked (DACP) | Etafilcon A, Pd 1 Masked, Pd 2 Unmasked (1DAVM) | Etafilcon A, Pd 1 Masked, Pd 2 Unmasked (DACP) | Nelfilcon A, Pd 1 Masked (1DAVM), Pd 2 Partial | Nelfilcon A, Pd 1 Masked (DACP), Pd 2 Partial | Etafilcon A, Pd 1 Masked (1DAVM), Pd 2 Partial | Etafilcon A, Pd 1 Masked (DACP), Pd 2 Partial | Nelfilcon A, Pd 1 Masked, Pd 2 Partial (1DAVM) | Nelfilcon A, Pd 1 Masked, Pd 2 Partial (DACP) | Etafilcon A, Pd 1 Masked, Pd 2 Partial (1DAVM) | Etafilcon A, Pd 1 Masked, Pd 2 Partial (DACP)
Number analyzed (Participants) | 23 | 23 | 28 | 28 | 23 | 23 | 28 | 28 | 20 | 20 | 25 | 25 | 20 | 20 | 25 | 25
Units on a scale | 94.1 (5.9) | 92.8 (6.5) | 94.1 (5.6) | 91.8 (6.4) | 93.7 (6.0) | 93.3 (5.7) | 95.2 (5.8) | 93.7 (6.6) | 93.4 (6.9) | 93.4 (7.1) | 93.6 (5.1) | 92.2 (5.6) | 92.3 (7.0) | 93.1 (7.0) | 93.5 (6.7) | 92.6 (5.8)
Statistical Analysis 1: Comparison: Nelfilcon A, Pd 1 Masked (1DAVM), Pd 2 Unmasked vs Nelfilcon A, Pd 1 Masked, Pd 2 Unmasked (1DAVM); Unmasked minus masked; Test type: Superiority or Other; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-2.2 to 1.4]
Statistical Analysis 2: Comparison: Nelfilcon A, Pd 1 Masked (DACP), Pd 2 Unmasked vs Nelfilcon A, Pd 1 Masked, Pd 2 Unmasked (DACP); Unmasked minus masked; Test type: Superiority or Other; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-1.5 to 2.5]
Statistical Analysis 3: Comparison: Etafilcon A, Pd 1 Masked (1DAVM), Pd 2 Unmasked vs Etafilcon A, Pd 1 Masked, Pd 2 Unmasked (1DAVM); Unmasked minus masked; Test type: Superiority or Other; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-0.1 to 2.2]
Statistical Analysis 4: Comparison: Etafilcon A, Pd 1 Masked (DACP), Pd 2 Unmasked vs Etafilcon A, Pd 1 Masked, Pd 2 Unmasked (DACP); Unmasked minus masked; Test type: Superiority or Other; Mean Difference (Final Values) = 1.9, 95% CI 2-sided [0.2 to 3.5]
Statistical Analysis 5: Comparison: Nelfilcon A, Pd 1 Masked (1DAVM), Pd 2 Partial vs Nelfilcon A, Pd 1 Masked, Pd 2 Partial (1DAVM); Partial masked minus masked; Test type: Superiority or Other; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.3 to 1.2]
Statistical Analysis 6: Comparison: Nelfilcon A, Pd 1 Masked (DACP), Pd 2 Partial vs Nelfilcon A, Pd 1 Masked, Pd 2 Partial (DACP); Partial masked minus masked; Test type: Superiority or Other; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.9 to 1.1]
Statistical Analysis 7: Comparison: Etafilcon A, Pd 1 Masked (1DAVM), Pd 2 Partial vs Etafilcon A, Pd 1 Masked, Pd 2 Partial (1DAVM); Partial masked minus masked; Test type: Superiority or Other; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-2.9 to 2.7]
Statistical Analysis 8: Comparison: Etafilcon A, Pd 1 Masked (DACP), Pd 2 Partial vs Etafilcon A, Pd 1 Masked, Pd 2 Partial (DACP); Partial masked minus masked; Test type: Superiority or Other; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-1.1 to 1.9]

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 03 May 2010 through 01 February 2011.
Description: This reporting group includes all enrolled and exposed participants.
Groups:
- Nelfilcon A: Nelfilcon A contact lenses
- Etafilcon A: Etafilcon A contact lenses
- 1DAVM: Etafilcon A with comfort additive contact lenses
- DACP: Nelfilcon A with comfort additive contact lenses
Arm/Group | Nelfilcon A | Etafilcon A | 1DAVM | DACP
Serious Adverse Events (participants affected / at risk) | 0/127 | 0/125 | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/127 | 0/125 | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
For a period of 10 years, the clinical investigator must hold all trial-related information and documents confidential and must agree to obtain sponsor's written consent before discussing, presenting, publicizing, or otherwise disclosing any preclinical and/or clinical data or impressions from this trial.